CLINICAL TRIAL: NCT04380649
Title: Brain Computer Interface Prototype Development for Assisted Alternative Communication in ALS
Brief Title: Development and Test of a Headset for BCI Until Obtaining an Efficient and Comfortable System That Can be Used in Daily Practice by ALS People
Acronym: TECH-ICOPA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-PP-18
Record Dates: First submitted 2020-04-22; First posted 2020-05-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Spinal Cord Diseases; Alternative Communication Devices; Neurodegenerative Diseases; Nervous System Diseases; Neuromuscular Diseases
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Spinal Cord Diseases; Neurodegenerative Diseases; Nervous System Diseases; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALS people with severe disability (Experimental)
  Interventions: Device: New headset prototype

INTERVENTIONS:
Device: New headset prototype — creation of a new headset prototype for using the P300 Speller, comfortable to use in everyday life by people with disabilities.

SUMMARY:
"Brain-computer interfaces (BCIs) are computer-based systems that acquire brain signals, analyze them, and translate them into commands that are relayed to an output device to carry out a desired action. BCIs represent a very active and promising field of research among devices for people with severe motor disabilities. As the currently available systems correspond to research prototypes, they are not adapted to daily live situations. On the other hand, some systems have recently been commercialized, principally for video games but they are not satisfactory for use as a substitute technology in disability.

A BCI's prototype for alternative communication using a virtual keyboard, the P300 Speller, has been developed by the National Institute for Research in Digital Science and Technology (Athena team - Nice University). This prototype includes an EEG-cap with gel based active electrodes. A recent study conducted on 20 patients with ALS (University Hospital, Nice) demonstrated the usability of the system and the patient satisfaction concerning the ease of use and utility. To achieve a system that can be used in daily live in severely disabled patients, technical developments are necessary.

The investigators have conceptualized and developed an ergonomic, comfortable, headset, including dry electrodes to allow a prolonged use of the system.

The purpose of the study conducted all along the development of the headset is to improve the developed system until a successful system is achieved. This study is a monocentric usability study conducted on ALS people.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years old
2. For women of childbearing potential, use of contraception for the duration of the study
3. Diagnosis of suspected ALS, possible, probable with ENMG, probable, defined according to the criteria of the World Federation of Neurology (revised El Escorial criteria, Airlie House Conference 1998)
4. Understanding of the objective of the study after describing the principle of the P300 Speller and the course of the study
5. Ability to follow the study procedure and to comply with the schedule of visits when entering the study
6. Expression of a P300 wave under the conditions of the study

Exclusion criteria

1. Psychiatric illness or dementia that may interfere with the patient's ability to follow study procedures
2. History of photosensitive epilepsy
3. Patient subject to protective measures
4. Non-correctable visual disturbances
5. Limited ability to concentrate.
6. Women who are pregnant or breastfeeding or who have planned a pregnancy during the course of the study.
7. Persons deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
prototype set-up time | at 6 months
  The time for setting up the prototype will be defined in seconds by the time elapsed between the start and stop of the stopwatch, the installation sequence being defined as follows:
  * start of the stopwatch: patient seated, equipment positioned on the table
  * patient or caregiver (depending on the patient's motor skills; 1 person): takes the prototype and positions it on the (patient's) skull
  * stopwatch stop: when the prototype is set up ready to operate
Quality of the impedance of each electrode | at 6 months
  The quality will be considered satisfactory if the impedance value of each of the electrodes is ≤ 1 000 kOhm, according to literature data.
Number of errors during calibration | at 6 months
  The number of errors in copying the 10 letters during the calibration phase will be counted.
Patient/caregiver satisfaction | at 6 months
  The evaluation of patient and caregiver satisfaction will be carried out using visual analogue scales (VAS rated from 0 to 10) on their feelings (patient/caregiver) of use.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Provence-Alpes-Côte d'Azur Region, France

IPD SHARING:
Plan to Share IPD: No